CLINICAL TRIAL: NCT04020133
Title: Analgesic Effect of Adding Popliteal Plexus Block to Standard Saphenous Nerve Block in Patients Scheduled for Elective Arthroscopic Anterior Cruciate Ligament Reconstruction : Randomized Observer Blind Clinical Trial
Brief Title: the Role of Popliteal Plexus Block in Pain Management After Anterior Cruciate Ligament Reconstruction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany M Yassin, MD, Associate professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D182
Record Dates: First submitted 2019-01-20; First posted 2019-07-15 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pain, Postoperative
Keywords: ACL; popliteal plexus block; saphenous nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (Active Comparator): this group will receive post-operative saphenous nerve block by 1mg/kg plain bupivacaine 0.5% plus epinephrine 0.05 mg.
  Interventions: Procedure: saphenous nerve block; Drug: Plain bupivacaine; Drug: 0.05 mg epinephrine
- the intervention group (Active Comparator): this group will receive popliteal plexus block by 1mg/kg plain bupivacaine 0.5% plus epinephrine 0.05 mg in addition to standard saphenous nerve block by 1mg/kg plain bupivacaine 0.5% plus epinephrine 0.05 mg.
  Interventions: Procedure: saphenous nerve block; Procedure: popliteal plexus block; Drug: Plain bupivacaine; Drug: 0.05 mg epinephrine

INTERVENTIONS:
Procedure: saphenous nerve block — The skin is disinfected and the saphenous nerve is located via Ultrasound . the transducer is placed anteromedially, approximately at mid-thigh level "a high-frequency linear probe 5Y12 MHz prepared in a sterile fashion" (Phillips HD11) .
  The block needle (Stimuplex; Braun Medical, Bethlehem, Pa), is inserted in plane in a lateral-to-medial orientation and advanced toward the femoral artery .Once the needle tip is visualized anterior to the artery and after careful aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection site . When injection of local anesthetic does not appear to result in its spread around the femoral artery, additional needle repositions and injections may be necessary.
  Other Names: adductor canal block
Procedure: popliteal plexus block — After doing saphenous nerve block , we will move distally with the artery in the adductor canal until it moves away from the sartorius muscle to enter adductor hiatus . here , we will inject L.A above artery and so , popliteal plexus block will be accomplished
  Arms: the intervention group
Drug: Plain bupivacaine — 15ml of plain bupivacaine 0.5% will be given in both blocks
Drug: 0.05 mg epinephrine — 0.05 mg epinephrine will be added to bupivacaine in both blocks to prolong their duration

SUMMARY:
Anterior cruciate ligament (ACL) injury is traumatic and debilitating and is typically repaired using an arthroscopic technique performed as an outpatient surgical procedure. However, many patients complain that the postoperative pain is severe for the first 48 hours following the ACL reconstruction .

Effective postoperative pain management is a critical component to recovery, effective rehabilitation and patient satisfaction. Following ACL reconstruction, psychological factors are predictive of outcomes, and pain levels are inversely associated with function and quality of life assessment.

ACL reconstruction procedures may reflect the complexity innervation of the anatomical areas involved, which includes the femoral nerve and its infrapatellar and saphenous branches, the obturator nerve, as well as the tibial and common peroneal branches of the sciatic nerve. Therefore, surgical variables, namely the location of surgical ports and the source of grafts used, and this creates challenge to anaesthesiologist to determine easy , safe and efficacious nerve block to be used in this setting .

A recently described popliteal plexus block(PPB) is claimed to anesthetize articular branches from the posterior obturator nerve and tibial nerve. It was recently confirmed in a cadaver study that injection of 10 mL of dye into the distal end of the adductor canal spreads via the adductor hiatus to the popliteal fossa and stains the popliteal plexus (PP).

A blockade of the popliteal plexus , has been claimed to produce an equivalent analgesic effect to sciatic nerve block after total knee arthroplasty without causing any motor weakness.

The current study hypothesize that combined saphenous nerve block with popliteal plexus block will enhance post operative analgesia after ACL reconstruction with motor sparing of thigh and leg muscles. Thus, faster recovery and earlier post-operative physiotherapy.

The objective of the current study is to evaluate analgesic effect of combined saphenous and popliteal plexus block as post -operative analgesia for anterior cruciate ligament reconstruction operation compared to standard saphenous nerve block .

Patients scheduled for ACL reconstruction will be randomly assigned into one of two groups: the intervention group will receive popliteal plexus block and saphenous nerve block and the control group will receive the standard saphenous nerve block only.

DETAILED DESCRIPTION:
This study will be performed in Fayoum university Hospital from january 2019 to january 2021 on 58 adult patients undergoing ACL operation after obtaining approval of the Scientific and Ethical Committee of El Fayoum University Hospitals, and written informed consent from the patients.

Randomization will be done by using computer-generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before the block. Neither the participants, the study investigators, the attending clinicians, nor the data collectors will be aware of groups' allocation until the study end. The Consolidated Standards of Reporting Trials (CONSORT) recommendations for reporting randomized, controlled clinical trials will be followed.

Preoperative preparation:

History taking , physical examination and investigations will be done according to the local protocol designed to evaluate the patients. which includes complete blood count, blood sugar level, serum urea and creatinine ,liver function tests,coagulation profile and electrocardiogram (ECG) Before surgery, the participants will receive education about the VAS pain score (0-100 mm) (where0=no pain and 100 = worst comprehendible pain)and the details of the nerve block procedures. After a 6 h fast, the patients will be taken into the operation theatre.

Intraoperative management :

The patient will receive Midazolam 0.03 mg/kg intravenous (IV) and Cefotaxime 1 gm as premedication . Monitors (pulse oximeter, electrocardiography and non invasive blood pressure ) will be applied.

Induction of general anaesthesia will be done via propofol 1-2 mg/kg , fentanyl 1-3 mic/kg and atracurium 0.5 mg/kg . Endotracheal tube will be inserted and the patient will be mechanically ventilated. Anesthesia will be maintained with oxygen and isoflurane 1-2 % or as required and atracurium 10mg every 30 minutes. Fentanyl boluses 0.5 μg/kg will be repeated if heart rate (HR) or mean arterial pressure (MAP) rise 20 % above baseline values . Ondansetron 4 mg IV dose will be administered for postoperative nausea and vomiting (PONV) prophylaxis 30 min before the end of the case; dexamethasone use will be avoided due to its potential confounding effect on the block characteristics.and then , nerve blocks will be given according to randomization.

The skin is disinfected and the saphenous nerve is located via Ultrasound . the transducer is placed anteromedially, approximately at mid-thigh level "a high-frequency linear probe 5Y12 megahertz (MHz) prepared in a sterile fashion" (Phillips HD11) . If the artery is not immediately obvious, several maneuvers can be used to identify it, including color Doppler scanning to trace the femoral artery caudally from the inguinal crease. Once the femoral artery has been identified, the probe is moved distally to trace the artery until it passes through the adductor hiatus to become the popliteal artery.

The block needle (Stimuplex; Braun Medical, Bethlehem, Pa), is inserted in plane in a lateral-to-medial orientation and advanced toward the femoral artery . the passage of the needle through the sartorius and/or adductor muscles and into the adductor canal is usually associated with a paresthesia in the saphenous nerve distribution. Once the needle tip is visualized anterior to the artery and after careful aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection site . When injection of local anesthetic does not appear to result in its spread around the femoral artery, additional needle repositions and injections may be necessary.

Then , moving distally with the artery in the adductor canal until it moves away from the sartorius muscle to enter adductor hiatus . here , L.A will be injected above the artery and so , popliteal plexus block will be accomplished .

Both blocks done via in injection 15 mg bupivacaine 0.5% + 0.05 mg epinephrine. After the block done , VAS score , BP , HR , cumulative and interval opioid consumption and sedation level via Ramsay sedation scale will be measured every 4 hours for 24 hours post-operatively .

Rescue analgesia in the form of morphine per a titration protocol (3 mg morphine sulfate IV as a bolus dose that could be repeated every 5 minutes with a maximum dose of 15mg per 4 hours or 45 mg per 24 hours) was employed if visual analog pain scale (VAS) > 4. The morphine titration protocol was suspended with Oxygen saturation < 95%; Respiratory rate < 10 / min; the development of sedation (Ramsay sedation scale >2); development of acute adverse effects (allergy, marked itching, excessive vomiting, and hypotension with systolic blood pressure _ 20% of baseline values); or attaining adequate level of analgesia.

Statistical Analysis:

Sample size was calculated using (G power version 3). Minimal sample size of patients was 26 in each group needed to get power level 0.80, alpha level 0.05 and 0.8 as an effect size in the time for painkiller request after the intervention between the two groups. To overcome problem of loss of follow up, calculated sample size was increased by 10% to reach 29 in each group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status I/II/III .
* Age > 18 years.
* Body mass index of <40 kg/m2 .

Exclusion Criteria:

* Patient refusal,
* Un-cooperative patients
* BMI>40kg/m2 .
* Allergy to local anaesthetics.
* Anticoagulation or bleeding disorders.
* Pre-existing peripheral neuropathies.
* Inflammation or infection over injection site.
* Daily morphine consumption > 40 mg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The duration of analgesia | 24 hours post-operative
  the pain will be assisted based on the time needed for the first dose rescue analgesia

SECONDARY OUTCOMES:
the cumulative opioid consumption | 24 hours post operative
  the total amount of opioid received post operative
The intervals between opioid (morphine) doses | 24 hours post-operative
  the time needed between two successive opioid doses
the quality of analgesia based on visual analogue scale (VAS) pain scores at rest | 4 hours post-operative
  Severity of pain estimated by visual analog score (VAS) (where 0 = no pain, and 100 = worst imaginable pain)
the quality of analgesia based on visual analogue scale (VAS) pain scores at rest | 8 hours post-operativE
  Severity of pain estimated by visual analog score (VAS) (where 0 = no pain, and 100 = worst imaginable pain)
the quality of analgesia based on visual analogue scale (VAS) pain scores at rest | 12 hours post-operative
  Severity of pain estimated by visual analog score (VAS) (where 0 = no pain, and 100 = worst imaginable pain)
the quality of analgesia based on visual analogue scale (VAS) pain scores at rest | 16 hours post-operative
  Severity of pain estimated by visual analog score (VAS) (where 0 = no pain, and 100 = worst imaginable pain)
the quality of analgesia based on visual analogue scale (VAS) pain scores at rest | 20 hours post-operative
  Severity of pain estimated by visual analog score (VAS) (where 0 = no pain, and 100 = worst imaginable pain)
the quality of analgesia based on visual analogue scale (VAS) pain scores at rest | 24 hours post-operative
  Severity of pain estimated by visual analog score (VAS) (where 0 = no pain, and 100 = worst imaginable pain)
Incidence of complications related to both techniques | 24 hours post-operatively
  complications related to the Block or drug administered
Incidence of nausea | 4 hours post-operative
  Morphine related side effect
Incidence of nausea | 8 hours post-operative
  Morphine related side effect
Incidence of nausea | 12 hours post-operative
  Morphine related side effect
Incidence of nausea | 24 hours post-operative
  Morphine related side effect
Incidence of vomiting | 4 hours post-operative
  Morphine related side effect
Incidence of vomiting | 8 hours post-operative
  Morphine related side effect
Incidence of vomiting | 12 hours post-operative
  Morphine related side effect
Incidence of vomiting | 24 hours post-operative
  Morphine related side effect
Incidence of pruritus | 4 hours post-operative
  Morphine related side effect
Incidence of pruritus | 8 hours post-operative
  Morphine related side effect
Incidence of pruritus | 12 hours post-operative
  Morphine related side effect
Incidence of pruritus | 24 hours post-operative
  Morphine related side effect
Rate of over-sedation | 4 hours post-operative
  Morphine related side effect
Rate of over-sedation | 8 hours post-operative
  Morphine related side effect
Rate of over-sedation | 12 hours post-operative
  Morphine related side effect
Rate of over-sedation | 24 hours post-operative
  Morphine related side effect
Incidence of urine retension | 4 hours post-operative
  Morphine related side effect
Incidence of urine retension | 8 hours post-operative
  Morphine related side effect
Incidence of urine retension | 12 hours post-operative
  Morphine related side effect
Incidence of urine retension | 24 hours post-operative
  Morphine related side effect
Patients satisfaction with postoperative analgesia | 24 hours post-operative
  Will be evaluated according to a satisfaction score (poor = 0; fair = 1; good = 2; excellent= 3)

CONTACTS AND LOCATIONS:
Overall Officials: Hany MO Yassin, MD, Principal Investigator — faculty of medicine , fayoum university
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Runge C, Moriggl B, Borglum J, Bendtsen TF. The Spread of Ultrasound-Guided Injectate From the Adductor Canal to the Genicular Branch of the Posterior Obturator Nerve and the Popliteal Plexus: A Cadaveric Study. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):725-730. doi: 10.1097/AAP.0000000000000675. PMID 28937534
- [Background] Runge C, Bjorn S, Jensen JM, Nielsen ND, Vase M, Holm C, Bendtsen TF. The analgesic effect of a popliteal plexus blockade after total knee arthroplasty: A feasibility study. Acta Anaesthesiol Scand. 2018 Sep;62(8):1127-1132. doi: 10.1111/aas.13145. Epub 2018 May 24. PMID 29797704
- [Background] Sehmbi H, Brull R, Shah UJ, El-Boghdadly K, Nguyen D, Joshi GP, Abdallah FW. Evidence Basis for Regional Anesthesia in Ambulatory Arthroscopic Knee Surgery and Anterior Cruciate Ligament Reconstruction: Part II: Adductor Canal Nerve Block-A Systematic Review and Meta-analysis. Anesth Analg. 2019 Feb;128(2):223-238. doi: 10.1213/ANE.0000000000002570. PMID 29064877
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Derived] Mahmoud A, Boules M, Botros J, Mostafa M, Ragab S, Alsaeid M. Analgesic Impact of a Popliteal Plexus Block to Standard Adductor Canal Block in Arthroscopic Anterior Cruciate Ligament Reconstruction: A Randomized Blind Clinical Trial. Pain Res Manag. 2021 Dec 17;2021:1723471. doi: 10.1155/2021/1723471. eCollection 2021. PMID 34956430